CLINICAL TRIAL: NCT01880723
Title: Modifying Genes in Cystic Fibrosis: The Beta-2 Adrenergic Receptors and Epithelial Na+ Channels
Brief Title: Utilizing Exhaled Breathe Condensate Collection to Study Ion Regulation in Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Courtney Wheatley, Graduate Research Assistant, University of Arizona
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 08-1123-01; 1R01HL108962-01 (NIH)
Record Dates: First submitted 2013-06-15; First posted 2013-06-19 (Estimated); Results first posted 2014-06-25 (Estimated); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Cystic Fibrosis; Healthy
Keywords: exhaled breath condensate; diffusion capacity of the lungs for carbon monoxide and nitric oxide; albuterol; peripheral oxygen saturation; ion regulation
MeSH Terms: conditions — Cystic Fibrosis | interventions — Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Albuterol (Experimental): 2.5 mg diluted in 3mL normal saline nebulized using a Power Neb2 nebulizer
  Interventions: Drug: Albuterol
- Saline (healthy only) (Placebo Comparator): nebulized 3 ml normal saline using a Power Neb2 nebulizer
  Interventions: Drug: Placebo saline

INTERVENTIONS:
Drug: Albuterol — 2.5 mg diluted in 3mL normal saline nebulized using a Power Neb2 nebulizer
  Arms: Albuterol
Drug: Placebo saline — nebulized 3mL normal saline) using a Power Neb2 nebulizer
  Arms: Saline (healthy only)

SUMMARY:
Our aims were to determine if exhaled breath condensate (EBC) could detect differences in ion regulation between cystic fibrosis (CF) and healthy and measure the effect of the albuterol on EBC ions in these populations. We hypothesized EBC chloride and sodium would be lower in CF patients at baseline and that albuterol would decrease EBC sodium and increase EBC chloride.

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects:

* no cardiovascular abnormalities
* not overweight BMI>25
* 18-55 years of age

CF subjects:

* mild to moderate CF (FEV1>40% predicted)
* clinically diagnosed with positive sweat test (sweat Cl->60mmol/L)
* 10-55 years of age
* clinically stable

Exclusion Criteria:

Healthy subjects will be excluded if:

* If unable to consent for him/herself (cognitive impairment)
* Have a history or evidence of cardiovascular and/or pulmonary abnormalities.
* Have an abnormal 12-lead EKG
* Have an abnormal pulmonary function test
* Have a history of asthma
* Have a history of renal disease or estimated creatinine clearance < 55ml/min
* Women who are pregnant or planning to become pregnant during the study

CF subjects:

* If unable to consent for him/herself (cognitive impairment)
* Physically unable to perform exercise or breathing tests
* Have a history of renal disease or estimated creatinine clearance < 55ml/min
* Women who are pregnant or planning to become pregnant during the study.
* Have an abnormal 12-lead EKG
* Cystic Fibrosis related diabetes is uncontrolled
* Forced Expiratory Volume after 1 second (FEV1) is less than 40% predicted
* Have a history of joint disease
* Have history of pulmonary exacerbation within the last two weeks
* Experienced pulmonary hemorrhage within 6 months resulting in greater than 50cc of blood in the sputum
* not currently enrolled in any other research study

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2009-05; Primary Completion 2012-07 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wayne J Morgan, MD, Principal Investigator — Department of Pediatrics- Pulmonology, Allergy and Immunology, University of Arizona, Tucson, Arizona; Cori M Daines, MD, Principal Investigator — Department of Pediatrics- Pulmonology, Allergy and Immunology, University of Arizona, Tucson, Arizona; Eric M Snyder, PhD, Principal Investigator — Department of Pharmacy Practice and Science, University of Arizona, Tucson, Arizona; Hanna Phan, PharmD, Principal Investigator — Department of Pharmacy Practice and Science, University of Arizona, Tucson, Arizona; Asad Patanwalla, PharmD, Principal Investigator — Department of Pharmacy Practice and Science, University of Arizona, Tucson, Arizona
Locations (1):
- Department of Pharmacy Practice and Science, University of Arizona, Tucson, Arizona, Tucson, Arizona, United States

REFERENCES:
- [Result] Foxx-Lupo WT, Wheatley CM, Baker SE, Cassuto NA, Delamere NA, Snyder EM. Genetic variation of the alpha subunit of the epithelial Na+ channel influences exhaled Na+ in healthy humans. Respir Physiol Neurobiol. 2011 Dec 15;179(2-3):205-11. doi: 10.1016/j.resp.2011.08.008. Epub 2011 Aug 26. PMID 21889619
- [Result] Baker SE, Wheatley CM, Cassuto NA, Foxx-Lupo WT, Sprissler R, Snyder EM. Genetic variation of alphaENaC influences lung diffusion during exercise in humans. Respir Physiol Neurobiol. 2011 Dec 15;179(2-3):212-8. doi: 10.1016/j.resp.2011.08.007. Epub 2011 Aug 26. PMID 21893217
- [Result] Wheatley CM, Foxx-Lupo WT, Cassuto NA, Wong EC, Daines CL, Morgan WJ, Snyder EM. Impaired lung diffusing capacity for nitric oxide and alveolar-capillary membrane conductance results in oxygen desaturation during exercise in patients with cystic fibrosis. J Cyst Fibros. 2011 Jan;10(1):45-53. doi: 10.1016/j.jcf.2010.09.006. Epub 2010 Nov 2. PMID 21050829
- [Result] Traylor BR, Wheatley CM, Skrentny TT Jr, Foxx-Lupo WT, Phan H, Patanwala AE, Morgan WJ, Daines CL, Sprissler R, Snyder EM. Influence of genetic variation of the beta2-adrenergic receptor on lung diffusion in patients with cystic fibrosis. Pulm Pharmacol Ther. 2011 Oct;24(5):610-6. doi: 10.1016/j.pupt.2011.06.001. Epub 2011 Jun 15. PMID 21703359
- [Result] Snyder EM, Wong EC, Foxx-Lupo WT, Wheatley CM, Cassuto NA, Patanwala AE. Effects of an inhaled beta2-agonist on cardiovascular function and sympathetic activity in healthy subjects. Pharmacotherapy. 2011 Aug;31(8):748-56. doi: 10.1592/phco.31.8.748. PMID 21923601

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy: Healthy control subjects
- Cystic Fibrosis: Patients diagnosed with cystic fibrosis
Period: Overall Study
Arm/Group | Healthy | Cystic Fibrosis
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy | Cystic Fibrosis | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 25 (6) | 22 (8) | 24 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 8 | 12 | 20
Weight (kg) [Mean (Standard Deviation); unit: kg] | 64 (9) | 60 (9) | 62 (9)
Height (cm) [Mean (Standard Deviation); unit: cm] | 169 (8) | 166 (8) | 167 (8)
BMI (kg/m2) [Mean (Standard Deviation); unit: kg/m2] | 23 (3) | 22 (3) | 22 (3)
BSA (m2) [Mean (Standard Deviation); unit: m2] | 1.7 (0.1) | 1.7 (0.2) | 1.7 (0.1)
VO2 peak (% predicted) [Mean (Standard Deviation); unit: percent predicted] | 108 (35) | 54 (24) | 85 (39)

OUTCOME MEASURES:

1. Primary Outcome: Exhaled Sodium (mmol/L)
Description: We collected exhaled breath condensate (EBC) samples, with subjects breathing on a Jaeger EcoScreen for 20 minutes. EBC samples were collected in cystic fibrosis and healthy subjects before and 30-, 60-, and 90-minutes following albuterol administration.
Time Frame: up to 90-minutes post albuterol
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Healthy | Cystic Fibrosis
Number analyzed (Participants) | 16 | 16
mmol/L
  Baseline | 2.58 (1.51) | 2.24 (1.09)
  30 minutes post | 1.97 (0.58) | 2.11 (0.93)
  60 minutes post | 2.37 (0.94) | 1.73 (0.85)
  90 minutes post | 2.23 (1.34) | 1.86 (0.93)

2. Secondary Outcome: Diffusion Capacity of the Lungs for Carbon Monoxide
Description: Using the rebreathe technique the diffusion capacity of the lungs for carbon monoxide and nitric oxide were measured, and this allowed for the determination of alveolar-capillary membrane conductance and pulmonary capillary blood volume. These measurements were made at baseline and 30-, 60- and 90-minutes post albuterol administration in cystic fibrosis and healthy subjects.
Time Frame: baseline, 30-, 60- and 90-minutes post albuterol administration
Measure: Mean (Standard Deviation); unit: mL/min/mmHg
Arm/Group | Healthy | Cystic Fibrosis
Number analyzed (Participants) | 16 | 16
mL/min/mmHg
  Baseline | 21.5 (5.8) | 17.3 (4.4)
  30 minutes post | 21.6 (5.3) | 17.4 (4.3)
  60 minutes post | 21.6 (6.2) | 17.0 (4.4)
  90 minutes post | 21.2 (5.5) | 17.1 (4.9)

3. Secondary Outcome: Diffusion Capacity of the Lungs for Nitric Oxide
Description: as for outcome 2
Time Frame: baseline, 30-, 60- and 90-minutes post albuterol administration
Measure: Mean (Standard Deviation); unit: mL/min/mmHg
Arm/Group | Healthy | Cystic Fibrosis
Number analyzed (Participants) | 16 | 16
mL/min/mmHg
  Baseline | 70.3 (18.9) | 55.0 (15.0)
  30 minutes post | 70.8 (16.7) | 56.4 (15.0)
  60 minutes post | 72.1 (19.2) | 56.2 (16.6)
  90 minutes post | 73.0 (20.6) | 58.5 (17.8)

4. Primary Outcome: Net Exhaled Chloride
Description: The calculation of net chloride efflux was used to account for the paracellular reabsorption of Cl- that will follow the reabsorption of Na+ to maintain electroneutral ion flux. Thus, the net chloride efflux calculation used was the gross chloride concentration plus the absolute value of the percent change in sodium from baseline multiplied by the gross chloride concentration for each time point:
  Net Cl- efflux - [Cl- X-min post] + (([Na+ X-min post]-[Na+Baseline])/ [Na+Baseline]) x [Cl- X-min post])
Time Frame: baseline to 90 minutes post albuterol administration
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Healthy | Cystic Fibrosis
Number analyzed (Participants) | 16 | 16
mmol/L
  Baseline | 0.064 (0.05) | 0.037 (0.02)
  30 minutes post | 0.078 (0.143) | 0.048 (0.031)
  60 minutes post | 0.084 (0.073) | 0.057 (0.038)
  90 minutes post | 0.077 (0.06) | 0.050 (0.016)

5. Secondary Outcome: Peripheral Oxygen Saturation
Description: A finger pulse oximeter allowed for the measurement of peripheral oxygen saturation at baseline, 30-, 60- and 90-minutes post albuterol in cystic fibrosis and healthy subjects.
Time Frame: baseline, 30-, 60- and 90-minutes post albuterol
Measure: Mean (Standard Deviation); unit: percent of oxygenated hemoglobin
Arm/Group | Healthy | Cystic Fibrosis
Number analyzed (Participants) | 16 | 16
percent of oxygenated hemoglobin
  Baseline | 99 (1) | 98 (1)
  30 minutes post | 100 (0) | 98 (1)
  60 minutes post | 99 (1) | 98 (1)
  90 minutes post | 99 (1) | 99 (1)

ADVERSE EVENTS:
Time Frame: Within the study visit (~2 hours)
Arm/Group | Healthy | Cystic Fibrosis
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No